CLINICAL TRIAL: NCT02292875
Title: An Optional Follow-Up Study to Evaluate the Continued Efficacy of ToleroMune Grass in Grass Allergic Subjects Following Challenge With Grass Allergen in an Environmental Exposure Unit.
Brief Title: ToleroMune Grass Follow on Study
Status: Completed | Type: Observational
Sponsor: Circassia Limited (Industry)
Collaborators: Adiga Life Sciences, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TG002B
Record Dates: First submitted 2014-11-13; First posted 2014-11-17 (Estimated); Last update posted 2014-11-17 (Estimated); Status verified 2014-11

CONDITIONS: Rhinoconjunctivitis; Grass Allergy
Keywords: Grass Allergy; Rhinoconjunctivitis; Environmental Exposure Unit; Immunotherapy; ToleroMune Grass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- TG002 Subjects: Subjects previously randomised in study TG002

SUMMARY:
Grass pollen allergens are recognised as a major cause of allergic diseases in humans and animals. Worldwide, at least 40% of allergic patients are sensitised to grass pollen allergens and between 50-90% of hayfever or seasonal allergy sufferers are allergic to grass pollen. ToleroMune Grass is a novel, synthetic, allergen-derived peptide desensitising vaccine, currently being developed for the treatment of grass allergy.

The purpose of this optional observational follow-on study is to further evaluate rhinoconjunctivitis symptoms on exposure to Grass in the EEU among subjects who completed all dosing visits in study TG002 approximately two years after the start of treatment.

DETAILED DESCRIPTION:
This is a follow-up study to a multi-centre, randomised, double-blind, placebo controlled, parallel group clinical study (TG002) which evaluated the efficacy, safety and tolerability of three doses of ToleroMune Grass versus placebo in grass allergic subjects. Subjects who completed TG002 in calendar year 2012 will undergo a further single exposure to grass allergens in an EEU.

ELIGIBILITY:
Inclusion Criteria:

* Previously randomised into study TG002, and completed all treatment visits and PTC during calendar year 2012

Exclusion Criteria:

* "Partly controlled" and "uncontrolled" asthama
* History of anaphylaxis to grass allergen
* FEV1 <80% of predicted
* Treatment with beta-blockers, alpha-adrenoreceptor blockers, tranquilizers or psychoactuve drugs
* Symptoms of a clinically relevant illness
* Subjects who cannot tolerate allergen challenge in the EEU

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject previously randomised in study TG002 and completed all dosing visits and the PTC
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2014-04; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Total Rhinoconjunctivitis Symptom Scores | 32 months post first dose in TG002

SECONDARY OUTCOMES:
Grass Specific Immunoglobulin A (IgA) | 32 months post first dose in TG002
Grass Specific Immunoglobulin E (IgE) | 32 months post first dose in TG002
Grass Specific Immunoglobulin G Isotype 4 (IgG4) | 32 months post first dose in TG002
Skin Prick Weal Diameter | 32 months post first dose in TG002
Adverse Events | 32 months post first dose in TG002

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Kanata, Ontario
  - Kingston, Ontario

REFERENCES:
- [Derived] Ellis AK, Frankish CW, Armstrong K, Steacy L, Tenn MW, Pawsey S, Hafner RP. Persistence of the clinical effect of grass allergen peptide immunotherapy after the second and third grass pollen seasons. J Allergy Clin Immunol. 2020 Feb;145(2):610-618.e9. doi: 10.1016/j.jaci.2019.09.010. Epub 2019 Sep 27. PMID 31568796